CLINICAL TRIAL: NCT01530178
Title: Sitagliptin Dose Determination Study in Type 1 Diabetes
Brief Title: Sitagliptin Dose Determination Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Rubina Heptulla, Division Chief of Pediatric Endocrinology & Diabetes, Albert Einstein College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-246
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Results first posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part A (Active Comparator): Sitagliptin 25mg
  Interventions: Drug: Sitagliptin
- Part B (Active Comparator): Sitagliptin 50mg
  Interventions: Drug: Sitagliptin
- Part C (Active Comparator): Sitagliptin 100mg
  Interventions: Drug: Sitagliptin
- Part D (Placebo Comparator): Placebo oral tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sitagliptin — In each intervention arm the participant receives a different dose of sitagliptin.
  Other Names: Januvia
  Arms: Part A; Part B; Part C
Drug: Placebo Oral Tablet
  Arms: Part D

SUMMARY:
There are many recent advances in insulin treatment of type 1 diabetes, however after a meal sugars are always a concern. There is a drug sitagliptin (Januvia) which is FDA approved to treat people with type 2 diabetes which helps correct their glucoses (sugars) after meals. This study is going to test whether this drug can improve the after meal sugars in people with type 1 diabetes. To test this you will be given a test mixed meal and its effects on insulin, other hormones that affect blood glucose as well as your sugar will be measured by a series of blood tests. Insulin dose will be reduced by 20-50% to prevent low blood sugars which might occur because of food staying longer in the stomach than usual or due to the suppression of a hormone called glucagon which increases blood sugar. If you qualify you will be given sitagliptin (Januvia) 3 different times in 25 mg, 50 mg and 100mg dosages. You and the researchers will not know which dose you are taking at any single visit. A total of 30 people in which some will be children aged 13- 17 and others will be adults aged 18-30 will participate. Some will have had diabetes for over a year, others will be within 3 months of having been found to have type 1 diabetes. Furthermore, only 18-30 year people who are diagnosed with type 1 diabetes for a year or more will be studied initially (4 subjects) to establish safety data before younger subjects are enrolled into the study.

DETAILED DESCRIPTION:
Rationale: Sitagliptin has been extensively studied in patients with type 2 diabetes mellitus, but there are no documented studies in the literature to establish a safe and efficacious dose in type 1 diabetes mellitus. Our previous experience with exenatide, which is a GLP-1 agonist and also with similar end pharmacological effects as Sitagliptin and other related published studies suggest that to avoid immediate post-prandial hypoglycemia insulin dose needs to be reduced when patients administer glucagon suppressors in conjunction with insulin. Hence, the dose of insulin will be decreased by 20-50% when Sitagliptin will be administered.

Sitagliptin will be given in three different doses to T1DM subjects within 3 months of diagnosis and also in a group of subjects > 1 year of their diagnosis. A paired crossover design study aims to establish an effective glucose-lowering dose that will additionally minimize side effects. Furthermore, only 18-30 year old subjects who are diagnosed with T1DM for a year or more will be studied initially (4 subjects) to establish safety data before younger subjects are recruited into the study. The data will be un-blinded after the completion of the first two adult subjects in order to analyze preliminary data and also to reapply for funding. Data Safety Monitoring Board will meet before the initiation of the study and before children are enrolled into the study. The safety data after the meeting will be submitted to the IRB for review.

Specific Aim: To establish a safe and an effective glucose-lowering dose of Sitagliptin in type 1 diabetes (T1DM) when used along with rapid acting insulin which will normalize post-prandial hyperglycemia and reduce hyper-glucagonemia and delay gastric emptying.

Hypothesis: A dose-response effect of Sitagliptin will be observed on gastric emptying and glucagon suppression in both new and established subjects with T1DM.

Study Design: Following informed consent (and with appropriate subject assent), each subject with TIDM will undergo 5 study visits: Screening, Part A (Sitagliptin 25 mg), Part B (Sitagliptin 50 mg), Part C (Sitagliptin 100 mg), and Part D (Placebo). A randomized double-blinded trial with a 4-period crossover design will be used to establish an ideal Sitagliptin dose for the adult age group (18-30 years). The adult study subject's and the study staff (except one person) will be blinded to the dose of Sitagliptin and they will do all the study Parts A, B, C and D in random order.

Montefiore Medical Center (MMC) Investigational pharmacy and one of the study staff (excluding the PI) will be un-blinded to the protocol for doing the randomization table, dispensing, checking the dose of study medication and scheduling the study visits (done by the study staff person). For the pediatric age group (13-17 years) it will be single blinded trial with single ascending dose sequential study. Pediatric study subject's will be blinded to the dose of Sitagliptin and they all will start with the placebo part and then proceed with the study parts with Sitagliptin 25 mg, 50 mg and 100 mg dose in a sequential order. The participants will be admitted to the CRC on four occasions for the Parts A, B, C and D and each admission will be 3-4 weeks apart.

Inclusion/ Exclusion Criteria Subjects with T1DM in the age group of 12-30 years without any concomitant illnesses except treated hypothyroidism will be recruited and also have an HbA1C less than 9 %. Menstruating women must have a negative pregnancy test. Lactating and pregnant women will be excluded and anyone with anemia defined by Hemoglobin of less than 12 gm/dl. Also, subjects with a history of substance abuse (evaluated by medical history and CRAFFT questionnaire which will be administered at the screening visit) will be excluded. The subject's should not be on any other medication which affects blood sugars.

Screening: After signing a consent form, a screening evaluation will be performed up to 28 days prior to study enrollment in the CRC for the Parts A, B, C or D. The evaluation will consist of medical history, physical examination (including height, weight, vital signs and tanner staging), and blood samples for clinical laboratory tests: CBC, LFTs, amylase, lipase, creatinine and HbA1C. The approximate volume of blood drawn is expected to be 12 ml. CRAFFT questionnaire will be administered. Also each subject will have a Dexcom™ Continuous Glucose Monitoring System inserted. It has three parts - a glucose sensor that is inserted subcutaneously, a transmitter which connects to the sensor electrode and is attached to the body and a receiver which displays the glucose values. It gets updated every 5 minutes. The subject will need to wear it for 7 days. Also, they will be asked to keep a log on diet, insulin and exercise while wearing the CGMS. We will try to schedule the next visit with in the 7 day period while they are on the CGMS so that they are admitted while their glucose levels are relatively stable. We will give an extra sensor with instructions on how to wear it in case they cannot come to the next visit with in the week.

Part A: The subjects will be admitted into the CRC around 6:30 AM. Vitals will be taken. IV will be placed and blood will be drawn to measure Stat CBC, HbA1C, Liver function tests, Serum Amylase, Serum Lipase and Serum Creatinine. Study will be continued only if their Hemoglobin is greater than 12 gm/ dl. Urine pregnancy test will be done for all female subjects prior to study. Insulin infusion through the subcutaneous pump will be continued or long acting analog, glargine will be given as per home regimen.

BLOOD SAMPLING AND MEDICATIONS: At approximately 0700 baseline blood samples will be drawn prior to study start for: glucose, insulin, glucagon, GLP-1, DPP-4 activity and Sitagliptin. Also, there will be blood draws at the following time points: -240 min, -180 min, -60 min, 0 min, 4 hrs. prior to the mixed meal and at 10, 20, 30, 40, 60, 90, 120, 150, 180, 210, 240, 360 min after. The insulin pump basal rate (or glargine) will be set to continue as per home regimen. Sitagliptin 25 mg will be administered at this point. At around 1100 (0 min), the pre-breakfast insulin bolus of rapid acting insulin will be given at 0 min. The insulin dose will be based on the patient's usual insulin to carbohydrate ratio. This dose will be reduced by 20-50% and the subject will be offered a standard liquid meal of Boost High Protein Drink, 12 Oz. (360 calories, 50 g of carbohydrates and 12 g of fat) and asked to consume it within a 10-15 minute period. This will be enriched with 1 gram of [1- 13C] glucose. Expired 13CO2 will be determined in breath at -240, 0, 10, 20, 30, 40 60, 90, 120, 150, 180, 210, 240, 360 min. Lunch will be provided after 240 min and an insulin bolus of rapid acting insulin will be given through the insulin pump (calculated according to subject's insulin to carbohydrate ratio and sensitivity factor) or through an insulin injection. They will stay for 2 more hours for the 360 min blood draw. Blood glucose concentrations will be measured at the bedside using an Analox glucose analyzer. Sitagliptin being a 24 hr medication pk data will be obtained at 0 and 360 min. For safety reasons the subject's will be put on a Dexcom CGMS and they will wear for a week. During this period they will keep a log sheet in which they will note the blood glucose, food and exercise activity. They will return that using a prepaid envelope which will be provided. The subject will be discharged after this. They will not be paid separately for transportation, parking or child care. A social security number will be required. It will be kept confidential. For minors, compensation will be given to the parent, but it is intended for the child.

A subject will be withdrawn from participating in the study if he/she meets any of the following conditions: 1) develops a chronic disease 2) develops anemia 3) becomes pregnant 4) develops a weight loss of greater than 10 pounds for unspecified reasons 5) loss of contact- if we are unable to reach a study subject (within 2 months of screening or completion of the first study) by phone or mail to schedule the next appointment. All study subjects (that are withdrawn from the study) will receive a phone call and a letter notifying them that they have been withdrawn. Blood samples will be kept for 20 years because some of the assays have not been developed for some of the hormone analyses. Since it is difficult to perform clinical studies in pediatrics, we feel it is better to bank blood samples and perform hormone analyses as newer assays become available rather than repeating the study.

Treatment of Hypoglycemia: If blood glucose values in a subject are less than 55 mg/dl, IV glucose of 5-10gm, or if blood glucose less than 50 mg/dl, 10-15 g will be administered for countering low blood glucose to achieve euglycemia (90-130 mg/dl). 1-2 doses of IV glucose should correct hypoglycemia. If more than 3-4 doses are required to achieve euglycemia, the study will be terminated and the subjects will be offered a meal tray and blood sugar rechecked to ensure euglycemia. After the completion of the first 2 study subjects, the data safety and monitoring committee will assess safety of the protocol, as well as drug doses and adjustments to the protocol will be made. If hypoglycemia occurs even with the reduced dose of insulin, further reduction in insulin dose will be advised. The total blood draw volume will be 175.4 cc (3/4 cup) for Part A, B, C and 121.4 cc (1/2 cup) for Part D.

Each study will be 3-4 weeks apart. Prior to each part, hemoglobin must be >12 g/dl and a female subject should test negative for pregnancy. Part B: Will be identical as part A except that Sitagliptin dose will be 50 mg. Part C: Will be identical as part A except that Sitagliptin dose will be 100 mg. Part D: Will be identical as part A except that the study subject will receive a placebo. In all the Parts B, C, D urine pregnancy test will be done before the visit for all female subjects. Also after each Part A, B, C, D the subject will be on Dexcom™ Continuous Glucose Monitoring System for 7 days and after that they will send that back to us using a prepaid mailing envelope.

Statistical Analysis Power Calculation: Data from an earlier trial determined that the mean area under the curve (AUC) for children with T1DM with insulin alone was 470 mg*hr/dl. The current trial is designed to detect a 20% difference in mean AUC for glucose in the 300 min period to 376 mg*hr/dl. In our previous study, r > 0.7 was noted between repeated measures (in same subjects) and that the standard deviation for our excursion measure AUC is approximately 30%. With these specifications the necessary sample size is 11 subjects. With a 40% drop out rate we would need a total of 15 subjects with TIDM. Power calculations were based on an alpha of 0.5 and power of 80% and two-tailed test. To stratify them in to recent onset Vs established onset we will recruit 15 of each (n = 30). Data Analysis: Blood glucose levels will be measured and AUC will be determined for glucose for a 300 min time period for all 4 studies and a two-tailed, repeated measures analysis of variance will be performed. A modified paired t-test will be used for post hoc multiple comparison. Regression analysis will be used to calculate a dose response curve for each individual and the hypothesis will hold true at a significance of 0.05. Similar analysis will also be carried out for insulin and glucagon. The pharmacokinetics of Sitagliptin will be analyzed by model dependent and model-independent means. AUC, plasma clearance, half-life and steady state volumes of distributions will be among the parameters determined. Pharmacokinetic data will be analyzed using ADAPT II software. The initial curve fits will be performed with the weighted least squares algorithm. Other strategies will be invoked as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 13 to 30 years
2. Subjects must be otherwise healthy except for T1DM, and treated for hypothyroidism if present
3. Menstruating women must have negative pregnancy test.
4. Hemoglobin (Hb) more than 12 g/dl

Exclusion Criteria:

1. Having any other chronic condition except hypothyroidism stable on medications
2. On chronic medications that may affect glucose excursions
3. Hemoglobin less than 12 g/dl
4. Positive pregnancy test (based on Urine)
5. Pregnant or lactating mothers
6. Known allergy to Januvia

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Heptulla, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine CRC, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 participants were screened. 2 did not meet the criteria. Patients were recruited from diabetes clinics, via fliers, and online postings on clinical trial sites.
Pre-assignment Details: Only 2 subjects underwent the study visit using sitagliptin 25mg. As we did not see a significant difference between the doses of 25 mg and 50 mg of Sitagliptin, we therefore continued the study visits for other subjects using only 50 mg and 100 mg of sitagliptin
Groups:
- Placebo/Sitagliptin 25mg/Sitagliptin 50mg/Sitagliptin 100 mg: Each of the two study subjects underwent four study visits, three to four weeks apart; at each visit receiving either placebo, Sitagliptin 25 mg, Sitagliptin 50mg, or Sitagliptin 100mg.
- Placebo/Sitagliptin 50mg/Sitagliptin 100 mg: Each of the six study subjects underwent three study visits, three to four weeks apart; at each visit receiving either placebo, Sitagliptin 50mg, or Sitagliptin 100mg.
Period: Overall Study
Arm/Group | Placebo/Sitagliptin 25mg/Sitagliptin 50mg/Sitagliptin 100 mg | Placebo/Sitagliptin 50mg/Sitagliptin 100 mg
Started | 2 | 6
Completed | 2 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Sitagliptin 25mg/Sitagliptin 50mg/Sitagliptin 100 mg | Placebo/Sitagliptin 50mg/Sitagliptin 100 mg | Total
Number analyzed (Participants) | 2 | 6 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (2.0) | 23.6 (4.1) | 23.7 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Better Targeted Blood Glucose Levels
Description: The current trial is designed to detect a significant difference in the mean glucose levels in the treatment group
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Sitagliptin 25 mg: Only two out of eight study subjects underwent four study visits, three to four weeks apart; at each visit receiving either Sitagliptin 25 mg, sitagliptin 50mg, sitagliptin 100mg or Placebo
- Sitagliptin 50 mg; Sitagliptin 100 mg: Each of the eight study subjects underwent three study visits, three to four weeks apart; at each visit receiving either Sitagliptin 25mg, sitagliptin 50mg, sitagliptin 100mg, or placebo
- Placebo: Each of the eight study subjects were treated with placebo
Arm/Group | Sitagliptin 25 mg | Sitagliptin 50 mg | Sitagliptin 100 mg | Placebo
Number analyzed (Participants) | 2 | 8 | 8 | 8
mg/dl | 184.1 (28.3) | 179.4 (36.6) | 153.6 (22.4) | 181.5 (45.1)
Statistical Analysis 1: Comparison: Sitagliptin 100 mg vs Placebo; Test type: Other — Non-specified; p = 0.003, ANOVA; Mean Difference (Final Values) = -27.91, 95% CI 2-sided [-44.7 to -11.2]
Statistical Analysis 2: Comparison: Sitagliptin 50 mg vs Placebo; Test type: Other — Non-specified; p = 0.68, ANOVA; Mean Difference (Final Values) = -2.131, 95% CI 2-sided [-12.91 to 8.652]
Statistical Analysis 3: Comparison: Sitagliptin 50 mg vs Sitagliptin 100 mg; Test type: Other; p = 0.0005, ANOVA; Mean Difference (Final Values) = -25.78, 95% CI 2-sided [-38.39 to -13.17]

ADVERSE EVENTS:
Time Frame: The adverse event data was collected over a period of 1 year.
Groups:
- Sitagliptin 25 mg: Each of the two study subjects underwent three study visits, three to four weeks apart; at each visit receiving either placebo, sitagliptin 50mg, or sitagliptin 100mg
- Sitagliptin 50 mg; Sitagliptin 100 mg; Placebo: Each of the eight study subjects underwent three study visits, three to four weeks apart; at each visit receiving either placebo, sitagliptin 50mg, or sitagliptin 100mg
Arm/Group | Sitagliptin 25 mg | Sitagliptin 50 mg | Sitagliptin 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/2 | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No